CLINICAL TRIAL: NCT04839172
Title: Study of the Effect of Football Practice on Bone Remodeling.
Brief Title: Effect of Football on the Musculoskeletal System and Hormonal System
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: Villarreal CF (Unknown)
Responsible Party: Principal Investigator, Isabel Almodóvar Fernández, PhD, Cardenal Herrera University
Other Study IDs: CMOTC
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Regional Body Composition; Cortisol and Testosterone Levels
Keywords: Regional body composition; Testosterone; Cortisol
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dual-energy X-ray Absorptiometry (DXA) scan — Longitudinal changes in body composition are examined over four consecutive seasons (2017-2018, 2018-2019, 2019-2020, 2020-2021), four times per season in the following stages: start-preseason, start-season, mid-season and end-season.
  Other Names: Fasting blood samples

SUMMARY:
Several studies have shown that football practice regulates bone remodeling, producing an increase of bone mineral density and reducing the risk of fractures. Thus, the aim of this study is to evaluate the effect of football practice on the regulation of bone turnover in Spanish adult football players. Thanks to the collaboration agreement "Aula Endavant" the Villarreal CF participates as a collaborator in this Project. This agreement allows us to use their facilities and to analyze several football players' data.

DETAILED DESCRIPTION:
Several studies have shown that football practice regulates bone remodeling, producing an increase of bone mineral density and reducing the risk of fractures. These studies are mainly performed in adolescents and there are few results obtained from European adults subjects. Thus, the aim of this study is to evaluate the effect of football practice on the regulation of bone turnover in Spanish adult football players. Secondary objectives include: describing bone mineral density values, evaluating percentage of total lean mass and body fat, describing dietary and physical habits and analyzing blood tests of professional football players. As well as, they include updating the current state of knowledge of the influence of sports on bone. Thanks to the collaboration agreement "Aula Endavant" the Villarreal CF participates as a collaborator in this Project. This agreement allows us to use their facilities and to analyze several football players' data. In addition, different members of the club will directly participate as researchers during the development of this study.

One of the strengths of this study is that the data were obtained from two consecutive seasons of an elite soccer team.

One of the potential limitations that we have faced in this study is that in order to obtain a large sample, it is necessary to analyse the soccers from two consecutive seasons, which makes the study temporarily longer than desired.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* aged between 18 and 40 years
* who practice soccer for more than 6 hours / week from the age of 10 to the present.

Exclusion Criteria:

* play other elite sports than soccer
* play 6 or more hours of recreational sports per week
* smokers
* individuals with chronic cardiovascular diseases, hypo and hyperthyroidism, hypertension, rheumatoid arthritis and osteoarthritis

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: male professional soccer players playing in the top soccer championship in Spain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
to examine the evolution of total and regional body composition and cortisol and testosterone levels of Spanish elite soccer players during a soccer season | 3 years
  to examine the evolution of total and regional body composition and cortisol and testosterone levels of Spanish elite soccer players during a soccer season

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Muñoz Macho, MD, Study Chair — Medical Services of Villarreal CF SAD
Locations (1):
- Villarreal CF, Villarreal, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No